CLINICAL TRIAL: NCT02834585
Title: Follow-up of Recurrences of Limb Soft Tissue Sarcomas in Patients With Localized Disease: Performance of Ultrasound
Brief Title: Magnetic Resonance Imaging or Ultrasound in Soft Tissue Tumors (MUSTT)
Acronym: MUSTT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Genova (Other)
Responsible Party: Principal Investigator, Alberto Tagliafico, Assistant Professor, University of Genova
Other Study IDs: 223REG2014
Record Dates: First submitted 2016-07-13; First posted 2016-07-15 (Estimated); Last update posted 2016-07-15 (Estimated); Status verified 2016-07

CONDITIONS: Sarcoma; Soft Tissue Tumors; Ultrasound; Magnetic Resonance Imaging; Diagnostic Accuracy; Sensitivity; Specificity; Follow-up
MeSH Terms: conditions — Sarcoma; Soft Tissue Neoplasms; Hypersensitivity | interventions — High-Energy Shock Waves

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Ultrasound: Patients undergoing Ultrasound
  Interventions: Other: Ultrasound
- Magnetic Resonance Imaging: Patients undergoing Magnetic Resonance Imaging
  Interventions: Other: Ultrasound

INTERVENTIONS:
Other: Ultrasound

SUMMARY:
Adult soft tissue sarcomas (STS) are rare tumours with an estimated incidence averaging 5/100 000/year in Europe. The prognosis of soft tissue sarcomas is dominated by local recurrence and distant metastasis. A link seems to exist between local recurrence and overall survival. Local recurrence occurs in approximately 16-29% of STS of the limbs. A combination of resection and radiotherapy is the optimal treatment of primary tumours according to histological grade and surgical result. Modern imaging techniques such as ultrasound (US), magnetic resonance (MR) and computed tomography (CT) are normally used to rule-out a recurrence in patients operated on for STS. However, none of this technique is perfect and different advantages and drawbacks have to be considered in choosing one or another technique. In the past, US was used in tumour follow-up to detect tumour recurrences, however these studies didn't use high-resolution transducers and the timing of imaging respect to surgery was not defined. The recent advances in transducer technology improved the diagnostic capabilities of US.

For the evaluation of limbs soft-tissue masses, US is widely used as a first level modality. The reasons are that US is widely available, fast, easily repeatable and often more accessible than CT and MR Imaging. In addition, US equipped with high-frequency transducers have a spatial resolution that may be comparable or higher than that of MR Imaging and CT in the evaluation of superficial soft-tissues. US and MR Imaging are often not able to differentiate benign from malignant tumours, therefore several lesions detected with US or MR Imaging warrant biopsy. The clinical practice guidelines of the ESMO (European Society of Medical Oncology) published in 2010 found that there are no published data to indicate the optimal routine follow-up policy of surgically treated patients with localized disease. Moreover, it has not been demonstrated that, for limb sarcomas recurrences, MR Imaging is superior and cost-effective compared to US for the assessment of the primary site. Considering that surgically treated intermediate-/high-grade patient may be followed frequently, even every 3-4 months in the first 2-3 years and considering that performing US is easier than having MR Imaging, the purpose of this study is to evaluate the diagnostic performance of US in the detection of local recurrences of adults patients with soft tissue sarcomas of the limb.

DETAILED DESCRIPTION:
Adult soft tissue sarcomas (STS) are rare tumours with an estimated incidence averaging 5/100 000/year in Europe. The prognosis of soft tissue sarcomas is dominated by local recurrence and distant metastasis. A link seems to exist between local recurrence and overall survival. Local recurrence occurs in approximately 16-29% of STS of the limbs. A combination of resection and radiotherapy is the optimal treatment of primary tumours according to histological grade and surgical result. Modern imaging techniques such as ultrasound (US), magnetic resonance (MR) and computed tomography (CT) are normally used to rule-out a recurrence in patients operated on for STS. However, none of this technique is perfect and different advantages and drawbacks have to be considered in choosing one or another technique. In the past, US was used in tumour follow-up to detect tumour recurrences, however these studies didn't use high-resolution transducers and the timing of imaging respect to surgery was not defined. The recent advances in transducer technology improved the diagnostic capabilities of US.

For the evaluation of limbs soft-tissue masses, US is widely used as a first level modality. The reasons are that US is widely available, fast, easily repeatable and often more accessible than CT and MR Imaging. In addition, US equipped with high-frequency transducers have a spatial resolution that may be comparable or higher than that of MR Imaging and CT in the evaluation of superficial soft-tissues. US and MR Imaging are often not able to differentiate benign from malignant tumours, therefore several lesions detected with US or MR Imaging warrant biopsy. The clinical practice guidelines of the ESMO (European Society of Medical Oncology) published in 2010 found that there are no published data to indicate the optimal routine follow-up policy of surgically treated patients with localized disease. Moreover, it has not been demonstrated that, for limb sarcomas recurrences, MR Imaging is superior and cost-effective compared to US for the assessment of the primary site. Considering that surgically treated intermediate-/high-grade patient may be followed frequently, even every 3-4 months in the first 2-3 years and considering that performing US is easier than having MR Imaging, the purpose of this study is to evaluate the diagnostic performance of US in the detection of local recurrences of adults patients with soft tissue sarcomas of the limb.

The clinical practice guidelines of the ESMO (European Society of Medical Oncology) published in 2010 found that there are no published data to indicate the optimal routine follow-up policy of surgically treated patients with localized disease. Moreover, it has not been demonstrated that, for limb sarcomas recurrences, MR Imaging is superior and cost-effective compared to US for the assessment of the primary site. Considering that surgically treated intermediate-/high-grade patient may be followed frequently, even every 3-4 months in the first 2-3 years, if US is demonstrated to be non-inferior to MRI a great sparing of healthcare resources will be warranted. In addition, patients operated on for localized soft tissue sarcomas of the limb will be possibly followed-up with clinical examination and US instead of MR Imaging.

ELIGIBILITY:
Inclusion Criteria:

* Patients operated on for localized soft tissue sarcomas of the limb

Exclusion Criteria:

* Unable to understand or execute written informed consent
* Unable or unwilling to agree to follow-up during observation period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients operated on for localized soft tissue sarcomas of the limb
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2014-10; Primary Completion 2020-01 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of US in the detection of local recurrences | 4 years

CONTACTS AND LOCATIONS:
Locations (1):
- UNIGE, Genova, Genova, Italy

REFERENCES:
- [Result] Tagliafico A, Truini M, Spina B, Cambiaso P, Zaottini F, Bignotti B, Calabrese M, Derchi LE, Martinoli C. Follow-up of recurrences of limb soft tissue sarcomas in patients with localized disease: performance of ultrasound. Eur Radiol. 2015 Sep;25(9):2764-70. doi: 10.1007/s00330-015-3645-z. Epub 2015 Mar 21. PMID 25794664